CLINICAL TRIAL: NCT00708682
Title: A Phase 3, Open Label, Single Arm Trial Evaluating the Safety, Tolerability, and Immunogenicity of 13-Valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in Mexico
Brief Title: Study Evaluating 13-Valent Pneumococcal Conjugate Vaccine in Healthy Infants in Mexico
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3009
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Vaccines, Pneumococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine

SUMMARY:
The purpose of this study will be to evaluate safety, tolerability and immunogenicity of 13-valent pneumococcal vaccine in healthy infants given with routine pediatric vaccinations in Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2 month infants, available for entire study period and parent/legal guardian reachable by telephone
* Able to complete three blood draws during study
* At least 3.5 kg at enrollment

Exclusion Criteria:

* Previous vaccination (except Hepatitis, BCG), contraindication or allergic reaction to vaccines
* Immune deficiency, bleeding disorder or significant chronic medical condition

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (8):
- Mexico (8):
  - Guadalajara, Jalisco
  - Distrio Federal, Mexico
  - Morelia, Michoacán
  - Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - Oaxaca City, Oaxaca
  - Puebla City, Puebla
  - Mérida, Yucatán

REFERENCES:
- [Derived] Rodgers GL, Esposito S, Principi N, Gutierrez-Brito M, Diez-Domingo J, Pollard AJ, Snape MD, Martinon-Torres F, Gruber WC, Patterson S, Thompson A, Gurtman A, Paradiso P, Scott DA. Immune response to 13-valent pneumococcal conjugate vaccine with a reduced dosing schedule. Vaccine. 2013 Oct 1;31(42):4765-74. doi: 10.1016/j.vaccine.2013.08.009. Epub 2013 Aug 16. PMID 23965217

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) dose administered intramuscularly (IM) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose)
Period: Infant Series
Arm/Group | 13vPnC
Started | 225
Vaccinated Dose 1 | 223
Vaccinated Dose 2 | 214
Vaccinated Dose 3 | 194
Completed | 192
Not Completed | 33
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 1
Not completed — Parent/legal guardian request | 6
Not completed — Failed to return | 2
Not completed — Other | 19
Period: After Infant Series
Arm/Group | 13vPnC
Started | 192
Completed | 191
Not Completed | 1
Not completed — Parent/Legal Guardian Request | 1
Period: Toddler Dose
Arm/Group | 13vPnC
Started | 191
Completed | 183
Not Completed | 8
Not completed — Parent/Legal Guardian Request | 1
Not completed — Lost to Follow-up | 3
Not completed — Failed to Return | 4

BASELINE CHARACTERISTICS:
Arm/Group | 13vPnC
Number analyzed (Participants) | 225
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 116

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level Greater Than or Equal to (≥) 0.35 Micrograms Per Milliliter (Mcg/mL), 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥0.35mcg/mL, along with the corresponding 95 percent confidence interval (95% CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable 3-Dose Infant Immunogenicity population: eligible participants who received treatments as assigned at all 3 doses, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 171
Percentage of participants
  Common serotypes - serotype 4 | 100.0 [97.9 to 100.0]
  Common serotypes - serotype 6B | 97.7 [94.1 to 99.4]
  Common serotypes - serotype 9V | 98.2 [94.9 to 99.6]
  Common serotypes - serotype 14 | 98.8 [95.8 to 99.9]
  Common serotypes - serotype 18C | 98.8 [95.8 to 99.9]
  Common serotypes - serotype 19F | 98.2 [95.0 to 99.6]
  Common serotypes - serotype 23F | 92.9 [87.9 to 96.3]
  Additional serotypes - serotype 1 | 99.4 [96.8 to 100.0]
  Additional serotypes - serotype 3 | 94.1 [89.4 to 97.1]
  Additional serotypes - serotype 5 | 98.2 [95.0 to 99.6]
  Additional serotypes - serotype 6A | 98.8 [95.8 to 99.9]
  Additional serotypes - serotype 7F | 98.8 [95.8 to 99.9]
  Additional serotypes - serotype 19A | 99.4 [96.8 to 100.0]

2. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35mcg/mL, 1 Month After Dose 2 of the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥0.35mcg/mL, along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after dose 2 of the infant series (5 months of age)
Population: Evaluable 2-Dose Infant Immunogenicity population: eligible participants who received treatments as assigned at dose 1 and dose 2, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 195
Percentage of participants
  Common serotypes - serotype 4 | 100.0 [98.1 to 100.0]
  Common serotypes - serotype 6B | 80.9 [74.7 to 86.2]
  Common serotypes - serotype 9V | 95.9 [92.1 to 98.2]
  Common serotypes - serotype 14 | 99.0 [96.3 to 99.9]
  Common serotypes - serotype 18C | 93.3 [88.9 to 96.4]
  Common serotypes - serotype 19F | 98.5 [95.5 to 99.7]
  Common serotypes - serotype 23F | 77.9 [71.5 to 83.6]
  Additional serotypes - serotype 1 | 98.5 [95.6 to 99.7]
  Additional serotypes - serotype 3 | 96.4 [92.7 to 98.5]
  Additional serotypes - serotype 5 | 97.4 [94.1 to 99.2]
  Additional serotypes - serotype 6A | 94.9 [90.8 to 97.5]
  Additional serotypes - serotype 7F | 99.0 [96.3 to 99.9]
  Additional serotypes - serotype 19A | 99.5 [97.2 to 100.0]

3. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Concentration ≥0.35mcg/mL, 1 Month After the Toddler Dose
Description: as for outcome 2
Time Frame: 1 month after the toddler dose (13 months of age)
Population: Evaluable Toddler Immunogenicity population: eligible participants who received treatments as assigned at all 3 doses of the infant series and at the toddler dose, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 155
Percentage of participants
  Common serotypes - serotype 4 | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 6B | 99.4 [96.5 to 100.0]
  Common serotypes - serotype 9V | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 14 | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 18C | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 19F | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 23F | 99.4 [96.5 to 100.0]
  Additional serotypes - serotype 1 | 100.0 [97.6 to 100.0]
  Additional serotypes - serotype 3 | 96.7 [92.5 to 98.9]
  Additional serotypes - serotype 5 | 100.0 [97.6 to 100.0]
  Additional serotypes - serotype 6A | 100.0 [97.6 to 100.0]
  Additional serotypes - serotype 7F | 100.0 [97.6 to 100.0]
  Additional serotypes - serotype 19A | 100.0 [97.6 to 100.0]

4. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal IgG Antibody After Dose 2 of the Infant Series
Description: Antibody GMC for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. GMCs were calculated using all participants with available data for the specified blood draw.
Time Frame: Dose 2 of infant series (4 months of age)
Population: Evaluable 2-Dose Infant Immunogenicity population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 195
mcg/mL
  Common serotypes - serotype 4 | 3.54 [3.16 to 3.97]
  Common serotypes - serotype 6B | 0.84 [0.71 to 0.98]
  Common serotypes - serotype 9V | 1.82 [1.60 to 2.08]
  Common serotypes - serotype 14 | 5.54 [4.72 to 6.50]
  Common serotypes - serotype 18C | 1.80 [1.56 to 2.07]
  Common serotypes - serotype 19F | 4.14 [3.59 to 4.78]
  Common serotypes - serotype 23F | 0.84 [0.71 to 0.99]
  Additional serotypes - serotype 1 | 3.41 [3.00 to 3.89]
  Additional serotypes - serotype 3 | 1.11 [1.01 to 1.23]
  Additional serotypes - serotype 5 | 1.89 [1.67 to 2.13]
  Additional serotypes - serotype 6A | 1.86 [1.60 to 2.16]
  Additional serotypes - serotype 7F | 2.98 [2.70 to 3.29]
  Additional serotypes - serotype 19A | 3.52 [3.07 to 4.03]

5. Other Pre Specified Outcome: GMC for Serotype-specific Pneumococcal IgG Antibody After Dose 3 of the Infant Series
Description: Antibody GMC for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 7vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. GMCs were calculated using all participants with available data for the specified blood draw.
Time Frame: Dose 3 of infant series (6 months of age)
Population: Evaluable 3-Dose Infant Immunogenicity population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 171
mcg/mL
  Common serotypes - serotype 4 | 3.48 [3.12 to 3.88]
  Common serotypes - serotype 6B | 5.02 [4.27 to 5.90]
  Common serotypes - serotype 9V | 2.34 [2.11 to 2.60]
  Common serotypes - serotype 14 | 9.35 [8.07 to 10.82]
  Common serotypes - serotype 18C | 2.50 [2.23 to 2.81]
  Common serotypes - serotype 19F | 3.75 [3.28 to 4.29]
  Common serotypes - serotype 23F | 1.83 [1.55 to 2.17]
  Additional serotypes - serotype 1 | 4.23 [3.73 to 4.79]
  Additional serotypes - serotype 3 | 1.17 [1.03 to 1.33]
  Additional serotypes - serotype 5 | 3.11 [2.75 to 3.52]
  Additional serotypes - serotype 6A | 4.08 [3.56 to 4.68]
  Additional serotypes - serotype 7F | 3.71 [3.34 to 4.12]
  Additional serotypes - serotype 19A | 4.19 [3.71 to 4.74]

6. Other Pre Specified Outcome: GMC for Serotype-specific Pneumococcal IgG Antibody After the Toddler Dose
Description: Antibody GMC for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 7vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. GMCs were calculated using all participants with available data after the toddler dose and after the third dose of the infant series.
Time Frame: Toddler Dose (12 months of age)
Population: Evaluable Toddler Immunogenicity population subset where the number of participants analyzed (N) equals (=) those who had a valid and determinate assay result for antibody GMC at both the infant dose 3 and toddler dose.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 137
mcg/mL
  Common serotypes - serotype 4 | 5.10 [4.41 to 5.89]
  Common serotypes - serotype 6B | 15.41 [12.92 to 18.38]
  Common serotypes - serotype 9V | 3.76 [3.29 to 4.29]
  Common serotypes - serotype 14 | 10.62 [9.16 to 12.32]
  Common serotypes - serotype 18C | 3.93 [3.45 to 4.48]
  Common serotypes - serotype 19F | 11.33 [9.68 to 13.26]
  Common serotypes - serotype 23F | 5.70 [4.81 to 6.77]
  Additional serotypes - serotype 1 | 5.86 [5.08 to 6.75]
  Additional serotypes - serotype 3 | 1.62 [1.42 to 1.84]
  Additional serotypes - serotype 5 | 4.75 [4.18 to 5.40]
  Additional serotypes - serotype 6A | 11.64 [9.93 to 13.64]
  Additional serotypes - serotype 7F | 5.81 [5.18 to 6.51]
  Additional serotypes - serotype 19A | 8.95 [7.84 to 10.23]

7. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 1 (2 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0cm); Moderate (2.5 to 7.0cm); Severe (greater than [>] 7.0cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 1 of Infant Series (2 months of age)
Population: Safety population: All participants who received at least 1 dose of the study vaccine; Number of participants analyzed (N) = those reporting yes for at least 1 day or no for all days for any local reaction.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 214
Percentage of participants
  Tenderness: Any | 63.5
  Tenderness: Significant | 12.4
  Swelling: Any | 31.2
  Swelling: Mild | 25.1
  Swelling: Moderate | 11.9
  Swelling: Severe | 0
  Redness: Any | 33.8
  Redness: Mild | 27.9
  Redness: Moderate | 10.6
  Redness: Severe | 0

8. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 2 (4 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 to 2.0cm); Moderate (2.5 to 7.0cm); Severe (>7.0cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 2 of Infant Series (4 months of age)
Population: Safety population; Number of participants analyzed (N) = those reporting yes for at least 1 day or no for all days for any local reaction.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 196
Percentage of participants
  Tenderness: Any | 69.4
  Tenderness: Significant | 12.6
  Swelling: Any | 29.9
  Swelling: Mild | 20.0
  Swelling: Moderate | 13.3
  Swelling: Severe | 0
  Redness: Any | 28.9
  Redness: Mild | 19.5
  Redness: Moderate | 12.3
  Redness: Severe | 0

9. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 8
Time Frame: Within 4 days after dose 3 (6 months of age)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 168
Percentage of participants
  Tenderness: Any | 61.3
  Tenderness: Significant | 15.4
  Swelling: Any | 29.4
  Swelling: Mild | 19.0
  Swelling: Moderate | 14.6
  Swelling: Severe | 0
  Redness: Any | 31.8
  Redness: Mild | 20.9
  Redness: Moderate | 13.9
  Redness: Severe | 0

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Toddler Dose (12 Months of Age)
Description: as for outcome 8
Time Frame: Within 4 days after toddler dose (12 months of age)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 154
Percentage of participants
  Tenderness: Any | 43.7
  Tenderness: Significant | 3.8
  Swelling: Any | 21.3
  Swelling: Mild | 8.1
  Swelling: Moderate | 15.8
  Swelling: Severe | 0
  Redness: Any | 22.0
  Redness: Mild | 8.8
  Redness: Moderate | 15.7
  Redness: Severe | 0

11. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 1 (2 Months of Age)
Description: Systemic events (any fever ≥ 38 degrees Celsius [C], decreased appetite, irritability, increased sleep, and decreased sleep) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 1 of Infant Series (2 months of age)
Population: Safety population; Number of participants analyzed (N) = those reporting yes for at least 1 day or no for all days for any systemic event.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 217
Percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C | 7.0
  Fever >39 degrees C but ≤40 degrees C | 0
  Fever >40 degrees C | 0
  Decreased appetite | 31.0
  Irritability | 69.8
  Increased sleep | 37.2
  Decreased sleep | 32.8

12. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 2 (4 Months of Age)
Description: as for outcome 11
Time Frame: Within 4 days after dose 2 of Infant Series (4 months of age)
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 198
Percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C | 18.5
  Fever >39 degrees C but ≤40 degrees C | 0.6
  Fever >40 degrees C | 0
  Decreased appetite | 29.3
  Irritability | 62.2
  Increased sleep | 24.5
  Decreased sleep | 35.1

13. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 11
Time Frame: Within 4 days after dose 3 of Infant Series (6 months of age)
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 172
Percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C | 18.3
  Fever >39 degrees C but ≤40 degrees C | 2.2
  Fever >40 degrees C | 0
  Decreased appetite | 25.7
  Irritability | 63.2
  Increased sleep | 22.9
  Decreased sleep | 37.3

14. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Toddler Dose (12 Months of Age)
Description: as for outcome 11
Time Frame: Within 4 days after toddler dose (12 months of age)
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 162
Percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C | 23.0
  Fever >39 degrees C but ≤40 degrees C | 0
  Fever >40 degrees C | 0
  Decreased appetite | 33.8
  Irritability | 46.7
  Increased sleep | 17.9
  Decreased sleep | 22.0

ADVERSE EVENTS:
Time Frame: Baseline through 1 Month after last study vaccination (13 Months). Local reactions and systemic events assessed within 4 days of dose: Infant Series Dose 1=2 months of age; Dose 2=4 months of age; Dose 3=6 months of age; Toddler Dose=12 months of age.
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Infant Series 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5mL dose administered intramuscularly (IM) at 2, 4, and 6 months of age (infant series).
  Other Adverse Events (AEs) (non-serious events): the number affected (n) for non-systematic (non-solicited) Other Adverse Events n=79; systematic (solicited) Any Local Reaction n=154, 139, and 112 for Dose 1, 2,and 3 of infant series, respectively; systematic (solicited) Any Systemic Event n=182, 144, and 126 for Dose 1, 2,and 3 of infant series, respectively.
- After the Infant Series 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series); assessment 1 month after the infant series (7 months of age).
- Toddler Dose 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 mL dose administered IM at 12 months of age (toddler dose).
  Other AEs (non-serious events): the number affected (n) for non-systematic (non-solicited) Other AEs n=50; systematic (solicited) Any Local Reaction n=73; systematic (solicited) Any Systemic Event n=96.
Arm/Group | Infant Series 13vPnC | After the Infant Series 13vPnC | Toddler Dose 13vPnC
Serious Adverse Events (participants affected / at risk) | 3/223 | 3/223 | 2/191
Other Adverse Events (participants affected / at risk) | 182/223 | 3/223 | 96/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (N=223) | After the Infant Series 13vPnC (N=223) | Toddler Dose 13vPnC (N=191)
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Kawasaki's disease (Vascular disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Breath holding (Psychiatric disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Seizure anoxic (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infant Series 13vPnC (N=223) | After the Infant Series 13vPnC (N=223) | Toddler Dose 13vPnC (N=191)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 0 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 7
Pyrexia (General disorders) | 6 | 0 | 14
Vaccination site pain (General disorders) | 0 | 0 | 3
Vaccination site erythema (General disorders) | 0 | 0 | 2
Vaccination site swelling (General disorders) | 0 | 0 | 2
Irritability (General disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 33 | 0 | 8
Viral upper respiratory tract infection (Infections and infestations) | 11 | 0 | 0
Pharyngitis (Infections and infestations) | 7 | 0 | 1
Bronchiolitis (Infections and infestations) | 6 | 0 | 0
Viral rhinitis (Infections and infestations) | 5 | 0 | 0
Rhinitis (Infections and infestations) | 4 | 0 | 0
Viral pharyngitis (Infections and infestations) | 4 | 0 | 0
Influenza (Infections and infestations) | 3 | 0 | 4
Impetigo (Infections and infestations) | 2 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Pyoderma (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tenderness (any) (Skin and subcutaneous tissue disorders) | 134/211 | 0/0 | 66/151 — Infant Series Dose 1 and Toddler Dose; tenderness (any)=present at site of vaccination
Tenderness (any) (Skin and subcutaneous tissue disorders) | 136/196 | 0/0 | 0/0 — Infant Series Dose 2; tenderness (any)=present at site of vaccination
Tenderness (any) (Skin and subcutaneous tissue disorders) | 100/163 | 0/0 | 0/0 — Infant Series Dose 3; tenderness (any)=present at site of vaccination
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 25/202 | 0/0 | 5/132 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 23/183 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)=present and interfered with limb movement
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 22/143 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)=present and interfered with limb movement
Swelling (any) (Skin and subcutaneous tissue disorders) | 64/205 | 0/0 | 30/141 — Infant Series Dose 1 and Toddler Dose; swelling (any)=present at site of vaccination
Swelling (any) (Skin and subcutaneous tissue disorders) | 56/187 | 0/0 | 0/0 — Infant Series Dose 2; swelling (any)=present at site of vaccination
Swelling (any) (Skin and subcutaneous tissue disorders) | 45/153 | 0/0 | 0/0 — Infant Series Dose 3; swelling (any)=present at site of vaccination
Swelling (mild) (Skin and subcutaneous tissue disorders) | 51/203 | 0/0 | 11/136 — Infant Series Dose 1 and Toddler Dose; swelling (mild)=present at site of vaccination
Swelling (mild) (Skin and subcutaneous tissue disorders) | 37/185 | 0/0 | 0/0 — Infant Series Dose 2; swelling (mild)=present at site of vaccination
Swelling (mild) (Skin and subcutaneous tissue disorders) | 28/147 | 0/0 | 0/0 — Infant Series Dose 3; swelling (mild)=present at site of vaccination
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 24/201 | 0/0 | 22/139 — Infant Series Dose 1 and Toddler Dose; swelling (moderate)=present at site of vaccination
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 24/180 | 0/0 | 0/0 — Infant Series Dose 2; swelling (moderate)=present at site of vaccination
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 21/144 | 0/0 | 0/0 — Infant Series Dose 3; swelling (moderate)=present at site of vaccination
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/199 | 0/0 | 0/132 — Infant Series Dose 1 and Toddler Dose; swelling (severe)=present at site of vaccination
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/177 | 0/0 | 0/0 — Infant Series Dose 2; swelling (severe)=present at site of vaccination
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/138 | 0/0 | 0/0 — Infant Series Dose 3; swelling (severe)=present at site of vaccination
Redness (any) (Skin and subcutaneous tissue disorders) | 69/204 | 0/0 | 31/141 — Infant Series Dose 1 and Toddler Dose; redness (any)=present at site of vaccination
Redness (any) (Skin and subcutaneous tissue disorders) | 54/187 | 0/0 | 0/0 — Infant Series Dose 2; redness (any)=present at site of vaccination
Redness (any) (Skin and subcutaneous tissue disorders) | 49/154 | 0/0 | 0/0 — Infant Series Dose 3; redness (any)=present at site of vaccination
Redness (mild) (Skin and subcutaneous tissue disorders) | 57/204 | 0/0 | 12/136 — Infant Series Dose 1 and Toddler Dose; redness (mild)=present at site of vaccination
Redness (mild) (Skin and subcutaneous tissue disorders) | 36/185 | 0/0 | 0/0 — Infant Series Dose 2; redness (mild)=present at site of vaccination
Redness (mild) (Skin and subcutaneous tissue disorders) | 31/148 | 0/0 | 0/0 — Infant Series Dose 3; redness (mild)=present at site of vaccination
Redness (moderate) (Skin and subcutaneous tissue disorders) | 21/199 | 0/0 | 22/140 — Infant Series Dose 1 and Toddler Dose; redness (moderate)=present at site of vaccination
Redness (moderate) (Skin and subcutaneous tissue disorders) | 22/179 | 0/0 | 0/0 — Infant Series Dose 2; redness (moderate)=present at site of vaccination
Redness (moderate) (Skin and subcutaneous tissue disorders) | 20/144 | 0/0 | 0/0 — Infant Series Dose 3; redness (moderate)=present at site of vaccination
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/199 | 0/0 | 0/132 — Infant Series Dose 1 and Toddler Dose; redness (severe)=present at site of vaccination
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/177 | 0/0 | 0/0 — Infant Series Dose 2; redness (severe)=present at site of vaccination
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/138 | 0/0 | 0/0 — Infant Series Dose 3; redness (severe)=present at site of vaccination
Fever ≥38°C but ≤39°C (General disorders) | 14/199 | 0/0 | 32/139 — Infant Series Dose 1 and Toddler Dose; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 33/178 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 26/142 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38°C but ≤39°C
Fever >39°C but ≤40°C (General disorders) | 0/199 | 0/0 | 0/132 — Infant Series Dose 1 and Toddler Dose; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 1/175 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 3/138 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39°C but ≤40°C
Fever >40°C (General disorders) | 0/199 | 0/0 | 0/132 — Infant Series Dose 1 and Toddler Dose; Fever >40°C
Fever >40°C (General disorders) | 0/175 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40°C
Fever >40°C (General disorders) | 0/138 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40°C
Decreased appetite (General disorders) | 63/203 | 0/0 | 51/151 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 55/188 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 38/148 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 148/212 | 0/0 | 71/152 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 120/193 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 103/163 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 77/207 | 0/0 | 25/140 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 45/184 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 35/153 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 67/204 | 0/0 | 31/141 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 66/188 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 56/150 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.